CLINICAL TRIAL: NCT04686890
Title: Erector Spinae Plane Block for Nefrectomy
Brief Title: Comparison of Erector Spinae Plane Block and Intravenous Analgesic in Nefrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, Zehra Ipek ARSLAN, Associate Professor, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: KIA 2020/96
Record Dates: First submitted 2020-12-07; First posted 2020-12-29 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-03

CONDITIONS: Regional Anesthesia Morbidity; Nephrectomy
Keywords: nefrectomy; erector spinea plane block
MeSH Terms: interventions — Tramadol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- postoperative opiod (morphine) consumption (Active Comparator): patient-controlled analgesia (15 minutes. lock time, 2 ml bolus= total 1 mg morphine intravenously, limited to maximum 4 bolus / per hour )
  Interventions: Procedure: erector spinea plane block administered preoperative open nephrectomy; Procedure: intravenous analgesic ( 1 mg/kg tramadol + non-steroid antiinflamatuar paracetamol )drug + 10 mg.kg
- peroperative continuous opioid (remifentanil) consumption (Active Comparator): continuous remifentanil infusion was given during the whole procedure
  Interventions: Procedure: erector spinea plane block administered preoperative open nephrectomy; Procedure: intravenous analgesic ( 1 mg/kg tramadol + non-steroid antiinflamatuar paracetamol )drug + 10 mg.kg
- postoperative numerated rating scale (Active Comparator): at the 1, 3, 6, 12 and 24 th hour postoperatively - numerated rating scale score was evaluated and recoded as 0= no pain (better), 10: unbearable pain (worse)
  Interventions: Procedure: erector spinea plane block administered preoperative open nephrectomy; Procedure: intravenous analgesic ( 1 mg/kg tramadol + non-steroid antiinflamatuar paracetamol )drug + 10 mg.kg

INTERVENTIONS:
Procedure: erector spinea plane block administered preoperative open nephrectomy — erector spinae plane block applied in this group before open nephrectomy
Procedure: intravenous analgesic ( 1 mg/kg tramadol + non-steroid antiinflamatuar paracetamol )drug + 10 mg.kg — intarvenous analgesic administered in this group for analgesia end of the open nephrectomy

SUMMARY:
The efficacy of erector spinae plane block versus intravenous analgesics compared relate to the morphine consumptions

DETAILED DESCRIPTION:
Patients undergoing elective nefrectomy were enrolled. Patients divided into two groups with a sealed envelope technique to ESP+ pca morphine group or iv analgesic + pca morphine group. All patients will premedicated. then esp will applied to one group before surgery at the preoperative care unit by the same anesthesiologist. The other group will receive intravenous tramadol 1 mg/kg + NSAID 1 ampule + parol 10 mg/ kg + ondansetron 4 mg bolus. İntravenous morphine pca with a concentration of 0.5 mg/cc were applied. And administered 1 mg boluses every 15 minutes lock time and 4 hour limit as 4 mg arranged. An anesthesia nurse who is responsible of all pcas' in the hospital was recorded the variables of these patients in the service

ELIGIBILITY:
Inclusion Criteria:18-65 years age

* ASA I-II
* undergoing elective nephrectomy

Exclusion Criteria:- ASA>3

* heart disease
* pregnancy
* lung disease
* scoliosis
* bleeding disorder
* infection at the manipulation side

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2020-12-30 (Actual); Primary Completion 2021-03-10 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Postoperative intravenous morphine patient controlled analgesia consumption | during postoperatively
  morphine consumptions were recorded till 24 th hour postoperatively
Peroperative remifentanyl consumption | Peroperatively
  Amount of Remifentanyl consumption recorded

SECONDARY OUTCOMES:
Visual analog rating scores | during postoperative surgery
  pain scores were recorded during surgery

CONTACTS AND LOCATIONS:
Overall Officials: Zehra Arslan, Principal Investigator — Kocaeli University Medical Faculty
Locations (1):
- Kocaeli University Medical Faculty, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No